CLINICAL TRIAL: NCT04301297
Title: Renal Manifestations of IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Faiza Kamal Abd Elkhalek, AssiutU, Assiut University
Other Study IDs: Renal manifestations of IBD
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To detect whether patients with inflammarory bowel disease (IBD) have some degree of renal involvement and also to determine if associated with disease activity or not.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) comprise two types of chronic intestinal disorders: Crohn's disease (CD) and ulcerative colitis (UC). CD involves the ileum and colon, but it can affect any region of the intestine, often discontinuously. UC involves the rectum and may affect part of the colon or the entire colon (pancolitis) in an un interrupted pattern. In Crohn's, the inflammation is often transmural, whereas in Ulcerative colitis the inflammation is typically confined to the mucosa . The extraintestinal manifestations of IBD are common and may occur in 25%-40% of patients. Inflammatory manifestations in the skin, eyes, liver and joints are considered primary manifestations. Development of primary extra intestinal manifestation appears to increase the risk of developing a second extra intestinal manifestation. Most IBD patients with extra intestinal manifestations have colonic inflammation, although some patients develop them prior to the onset of colonic symptoms. Extra intestinal manifestations are usually present at the time of active phase of IBD . In recent years, there have been reports on renal and urologic complications of IBD. They were mostly found to be related to ureteral obstruction by oxalate stones, cystitis, acute tubular necrosis due to volume depletion and AA amyloidosis. Nephrolithiasis and obstructive uropathy are especially seen with small bowel dysfunction. In a great proportion of IBD patients, ureteral obstruction is not caused by stones. This non calculus obstruction can occur in 50%-73% of CD patients and 50% of UC patients, and is usually caused by retroperitoneal local inflammation or by surgical complication (sutures) or colon cancer . There have also been reports of interstitial nephritis, mainly due to applied anti-inflammatory therapy, such as 5-aminosalicylic acid (5-ASA). Serious renal impairment is reported to occur in 1 of 500 patients treated with 5-ASA derivative. On the other hand, there are some reports that renal tubular damage is an extra intestinal manifestation of IBD and not a toxic side effect of anti-inflammatory therapy using 5-ASA or sulfasalazine. Furthermore, renal failure due to glomerulonephritis (GN) caused by the immune complex has been reported in several cases as an extraintestinal manifestation of IBD.

ELIGIBILITY:
Inclusion Criteria:

- A ny patients with IBD

Exclusion Criteria:

Pregnant kidney disease

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with IBD without any of exclusion criteria will be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Renal manifestations of IBD | 12 month
  Access renal manifestations of IBD

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Asyut, Egypt

REFERENCES:
- [Background] Ambruzs JM, Larsen CP. Renal Manifestations of Inflammatory Bowel Disease. Rheum Dis Clin North Am. 2018 Nov;44(4):699-714. doi: 10.1016/j.rdc.2018.06.007. Epub 2018 Sep 7. PMID 30274631